CLINICAL TRIAL: NCT02341196
Title: Randomized Clinical Trial of Polyester vs. Polyurethane Patch for Carotid Endarterectomy. Long-term Results
Brief Title: Randomized Clinical Trial of Polyester vs. Polyurethane Patch for Carotid Endarterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Poitiers (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBR01
Record Dates: First submitted 2014-12-21; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Carotid Artery Thrombosis; Carotid Artery Stenosis; Stroke
MeSH Terms: conditions — Carotid Artery Thrombosis; Carotid Stenosis; Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CEA + Polyester patch (Experimental): 225 Patients
  Interventions: Procedure: CEA
- CEA + Patch Polyurethane (Experimental): 225 Patients
  Interventions: Procedure: CEA

INTERVENTIONS:
Procedure: CEA — Patients in both groups received an intra-operative angiography
  Other Names: Carotid endarterectomy

SUMMARY:
This study examines the risk of thrombogenicity of the carotid patches in polyurethane compared to carotid patches in polyester including death, any stroke, carotid thrombosis at 30 days and long-term results including stroke and recurrent carotid stenosis at 10 years.

This study was run at the University of Roma, La Sapienza and at the University of Poitiers, randomisation was done in both enters after approval by the Ethical committee of the University of Roma (Record uploaded)

DETAILED DESCRIPTION:
This study examines the risk of thrombogenicity of the carotid patches in polyurethane compared to carotid patches in polyester including death, any stroke, carotid thrombosis at 30 days and long-term results including stroke and recurrent carotid stenosis at 10 years.

598 patients were considered for randomisation between January 1995 and January 2004. The following patients were excluded for randomisation (Redo carotid surgery: N=34, radiation induced carotid stenosis:N=45, indication for carotid bypass: N=65, Refusal of randomisation: N=4).

In total, 450 patients were randomized in two groups, 225 received a polyester patch and 225 received a polyurethane patch.

All patients were operated under general anaesthesia and all received an intraoperative angiography. A shunt was selectively used in patients with a recent stroke (<15 days) or with a contralateral carotid occlusion

ELIGIBILITY:
Inclusion Criteria:

* Carotid stenosis > 60% NASCET criteria

Exclusion Criteria:

* Redo carotid surgery
* Radiation induced carotid stenosis
* Extensive carotid lesion > 5 cm in length with involvement of the common carotid artery best treated by a carotid bypass

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 1995-01; Primary Completion 2004-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
carotid artery restenosis | 5 to 10 years after surgery
  Restenosis of carotid endarterectomy > 70% in diameter occurring 5 to 10 years after surgery diagnosed by color duplex ultrasound

SECONDARY OUTCOMES:
Any death occurring during follow-up | Time 0 (operation) to 10 years after surgery
  All death even those not related to carotid surgery
Any ipsilateral stroke | 0 days to 10 years
  Any paralysis occurring in relation with the operated carotid artery and lasting more than 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Illuminati, MD, PhD, Study Chair — University of Roma La Sapienza